CLINICAL TRIAL: NCT05141578
Title: Tailored, Multidomain, and Coach-assisted Interactive Mobile Application for the Adoption and Maintenance of a Healthy Lifestyle in Middle-aged and Older Adults With Modifiable Risk Factors for Dementia: A Pilot Feasibility Study
Brief Title: Multidomain Intervention on Modifiable Lifestyle Risk Factors for Dementia Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LuciLab (Industry)
Collaborators: Centre de Recherche de l'Institut Universitaire de Geriatrie de Montreal (Other); Sojecci II Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: LUCI-02
Record Dates: First submitted 2021-11-19; First posted 2021-12-02 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2021-12

CONDITIONS: Risk Behavior; Cognitive Decline
Keywords: Primary Prevention; Aging; Cognition
MeSH Terms: conditions — Risk-Taking; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Luci Intervention (Experimental): Participants enrolled in this group will receive the Luci intervention for a 24-week period.
  Interventions: Behavioral: Luci Coach Assisted Intervention
- Wait-list Control (No Intervention): Participants in the waiting-list control group will not receive any intervention during the study. They will be invited to participate to the program at the end of the trial.

INTERVENTIONS:
Behavioral: Luci Coach Assisted Intervention — The Luci intervention is a personalized behaviour change program delivered via an interactive mobile platform with the online support of a coach. It targets 3 lifestyle domains: physical activity, healthy diet and cognitive engagement.
  Participants in this group will be encouraged to adopt a healthy lifestyle, as a means for cognitive decline/dementia risk reduction. This will be achieved by providing educational materials, practical tips and strategies, and by assisting participants outlining goals to progressively adopt and maintain a healthier lifestyle.
  Coaching sessions will be held on a weekly basis from week 1 to 12, and every 2 weeks from week 13 to 24.
  Arms: Luci Intervention

SUMMARY:
The overarching aim is to develop and deploy a multidomain intervention delivered on a mobile application to help middle-aged to older adults reduce their risk for dementia by improving a set of modifiable lifestyle risk factors associated with cognitive decline/dementia. This registration concerns the Pilot Feasibility study which examines different aspects of feasibility in a small-scale randomized pilot study, before implementing an efficacy study on a larger sample. A secondary objective is to determine whether the program can result in a larger improvement on risk factors (measured with Behavioural Risk outcomes) compared to a control intervention. It is expected that persons enrolled in the Luci program show larger change in Behavioural Risk outcomes than those enrolled in the comparator condition.

DETAILED DESCRIPTION:
Multidomain lifestyle interventions show promising results in reducing the risk of cognitive decline and dementia.

In this study, we pilot the feasibility of a coach-based digital multidomain risk-reduction program to improve cognitive engagement, physical activity, and healthy eating in older adults at risk of dementia. This trial is the second step in the clinical validation process of the Luci program (see NCT04616794). In this 24-week study, participants are randomly assigned to the Luci Intervention group or to the Waiting-list Control group (i.e., participants receive the program after the end of the trial). Assessments will be done at study entry (T1), week 12 (T2), and week 24 (T3).

ELIGIBILITY:
Inclusion criteria:

* Proficient or native speakers in French;
* Computer literate defined as being able to read mails and browse the Internet, and having access to a computer, smartphone or tablet with an Internet connection;
* Committed not to participate in another program related to any of the three intervention domains for the duration of the trial;
* At least one of the following:

  * Low cognitive engagement in cognitively stimulating activities, defined as a score ≤ 22 on the adapted Cognitive Activity Questionnaire;
  * Low level of physical activity defined as less than 150 minutes/week) of moderate to vigorous physical activity measured using the Godin-Shephard Leisure Time Physical Activity Questionnaire, and no medical contraindication to physical activity based on the Physical Readiness Questionnaire for Everyone (PAR-Q+);
  * Low adherence to the Mediterranean-type diet defined as a score of ≤ 8 on the adapted Canadian Mediterranean Diet Scale, and no severe food allergy or intolerance or history of eating disorder.

Exclusion Criteria:

* Presence of a cognitive impairment as measured by the Cogstate Brief BatteryTM.
* General anesthesia within the last 6 months;
* Participation in any previous validation studies related to the program;
* Participation, currently or within the last 6 months, in a program where they received any of the three interventions;
* Unable to commit participation over the period of the study.
* Participants in the precontemplation stage of change.
* Participants with a high level of perceived stress;
* Having received a diagnosis of:

  * Dementia or neurodegenerative disease (AD and other dementias);
  * Past or present neurological disorder (multiple sclerosis, brain tumour, epilepsy, stroke, traumatic brain injury);
  * Severe psychiatric disorder (schizophrenia, major depression, bipolar disorder);
  * Uncontrolled cardiovascular or metabolic diseases;
  * Alcoholism or drug addiction;
  * Any other conditions expected to limit participation (e.g., visual acuity).

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2022-06-21 (Actual)

PRIMARY OUTCOMES:
Enrollment Ratio | At baseline post-enrollment
  Screening-to-enrollment ratio will be calculated as the number of enrolled participants over the number of screened participants.
Recruitment Rate | At baseline post-randomization
  Recruitment rate will be calculated as the number of participants randomized per month over the recruitment period
Acceptability of randomization | Week 24
  Acceptability of randomization will be assessed by comparing the post-randomization dropout rate in the control group relative to the intervention group.
Retention rate | Week 24
  Retention rate will be calculated as the proportion of randomized participants completing at least one of the measures at study end.
Program adherence | Week 24
  Program adherence will be calculated as the number of participants from the Luci condition who attend at least 66% of the prescribed coaching sessions over the 24-week intervention period.

SECONDARY OUTCOMES:
Change from baseline in Cognitive Engagement | At baseline, week 12, week 24
  Cognitive engagement is measured using the Cognitive Activity Questionnaire. Participants are asked to indicate the frequency in which they engage in 10 cognitive leisure activities. Scores range from 0 to 70. A higher score represents a higher cognitive engagement level.
Change from baseline in Physical Activity | At baseline, week 12, week 24
  Physical activity will be measured using the modified Godin-Shephard Leisure Time Physical Activity Questionnaire. An overall physical activity score is computed in Metabolic equivalent tasks (MET)-minutes/week, as well as a moderate-to-vigorous physical activity score. A higher MET value represents a higher physical activity level.
Change from baseline in Sitting Time | At baseline, week 12, week 24
  Sitting time will be investigated using a single question from the International Physical Activity Questionnaire. Participants will be asked the following question "During the last 7 days, how much time in total did you usually spend sitting on a week day?" (Number of hours and minutes, Don't know). A lower value represents a lower sitting time.
Change from baseline in Mediterranean Diet Adherence | At baseline, week 12, week 24
  Adherence to the Mediterranean Diet is measured with an adaptation of the Canadian Mediterranean Diet Scale. The scale consists of 13 questions on food consumption frequency and intake habits. Scores range from 0 to 13, where a higher score represents a higher adherence level.
Change from baseline in Luci Cognitive Engagement Score | At baseline, week 12, week 24
  Six questions are added to the Cognitive Activity Questionnaire to include activities not covered in the original questionnaire. All 16 items will be used to calculate the Luci Cognitive Engagement score. Scores range from 0 to 112. A higher score represents a higher cognitive engagement level.
Change from baseline in Luci Physical Activity Score | At baseline, week 12, week 24
  For 15 physical activity types, three questions will assess frequency, duration and intensity of activity on a typical week over the past 30 days. Responses will be used to calculate the Luci Physical Activity score as well as 3 subscores related to aerobic exercise, muscular resistance, and flexibility training, respectively. The total score and subscores are in Metabolic equivalent tasks (MET)-minutes/week. A higher score represents a higher physical activity level.
Change from baseline in Luci Medi Diet Adherence Score | At baseline, week 12, week 24
  Five questions are added to the Canadian Mediterranean Diet Scale to include food groups and food intake habits not covered in the original questionnaire. From the whole questionnaire, we selected 14 items that are most relevant for the intervention and grouped them into 12 categories to calculate the Luci Medi Diet adherence score. Scores range from 0 to 36, where a higher score represents a higher adherence level.
Goal Attainment (Luci Coach Assisted Intervention condition only) | On a weekly basis from week 1 to 12, and every 2 weeks from week 13 to 24
  Goal attainment will be self-rated by participants in the Luci Intervention group. For each goal, an indicator of perceived goal attainment will be established as well as an indicator of their perceived effort towards goal attainment. These will be reported using a 3-item categorical scale.
Perceived Progress | Week 12, week 24
  Perceived Progress domain specific will be rated on a 10-point Likert-scale.
Change from baseline in Readiness to Change (Luci Coach Assisted Intervention condition only) | At baseline, week 24
  Readiness to change will be determined using a 5-item categorical question.
Action Taken | At baseline, week 24
  Action taken will be measured using a 3-item question (Yes, No, Don't know).
Change from baseline in Expectation (Luci Coach Assisted Intervention condition only) | At baseline, week 24
  For each selected domain, participants' expectations will be assessed using a 7-point Likert scale.
Overall User Experience (Luci Coach Assisted Intervention condition only) | Week 24
  Different sets of measures will assess user experience. They will evaluate quality and usability of the platform, and participants' satisfaction and continuance usage intention of the program. Feedback about the overall user experience with the platform will be collected using a semi-structured interview conducted by phone.
Platform Usage | Continuously from baseline until week 24
  Continuous measures of different parameters linked to platform usage during the study period will be recorded and analyzed, including pattern of use (e.g., time of day), frequency (e.g., number of platform access), duration of use (e.g., duration of the coach sessions) and the functionalities used (e.g., content viewed).
Change from baseline in Cognitive Performance | At baseline, week 24
  Cognitive performance will be assessed using the Cogstate Brief Battery. Scores range from 0 to 200, where a score ≤ 90 will indicates a cognitive impairment.
Change from baseline in Current memory concerns | At baseline, week 24
  Memory concerns will be evaluated using 2 Yes/No questions.
Change from baseline in Perceived Stress | At baseline, week 24
  Perceived stress will be investigated using a 5-item categorical question, where a higher score indicates a higher stress level.
Change from baseline in Sleep Quality | At baseline, week 24
  Sleep quality will be assessed using a 4-point Likert scale, where a higher score indicates worse sleep quality.
Change from baseline in Depression | At baseline, week 24
  Depression will be assessed using a single Yes/No question.
Change from baseline in Quality of Life | At baseline, week 24
  Quality of life will be measured with the SF-12. Scores range from 0 to 100, where a higher score represents higher levels of quality of life.
Change from baseline in Dementia Literacy | At baseline, week 24
  Dementia literacy will be assessed using 20 questions. These will be answered using 5-point categorical scales.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Belleville, PhD, Principal Investigator — Centre de recherche de l'Institut Universitaire de gériatrie de Montréal
Locations (1):
- Lucilab, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No